CLINICAL TRIAL: NCT07279506
Title: Randomized Clinical Investigation Of The IXIUM TWIN Viscoelastic Ophthalmic Device (OVD) For Cataract Surgery With Intraocular Lens Implantation
Brief Title: Clinical Investigation of IXIUM TWIN Viscoelastic Ophthalmic Device For Cataract Surgery
Acronym: IXIUM_TWIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LCA Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024-A01718-39; 2024-A01718-39 (Other: ANSM)
Record Dates: First submitted 2025-11-24; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Cataract Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IXIUM TWIN (Experimental): IXIUM TWIN as the Ophthalmic Viscosurgical Devices in the cataract surgeryfor the cataract surgery
  Interventions: Device: IXIUM TWIN
- HEALON (Active Comparator): HEALON as the Ophthalmic Viscosurgical Devices in the cataract surgeryfor the cataract surgery
  Interventions: Device: HEALON

INTERVENTIONS:
Device: IXIUM TWIN — Use of IXIUM TWIN as the Ophthalmic Viscosurgical Devices in the cataract surgery
  Arms: IXIUM TWIN
Device: HEALON — Use of HEALON as the Ophthalmic Viscosurgical Devices in the cataract surgery
  Arms: HEALON

SUMMARY:
This clinical trial is testing a new surgical gel called IXIUM TWIN, designed to protect the eye during cataract surgery. Cataracts, which cloud the eye's natural lens, are the leading cause of vision loss worldwide. Surgery to remove the cataract and replace it with an artificial lens is the standard treatment, and viscoelastic gels like IXIUM TWIN are used to keep the eye stable and safe during the procedure.

The goal of this study is to compare IXIUM TWIN with an already approved gel (HEALON) to ensure it works just as well (or better) in protecting the delicate cells inside the eye. Specifically, researchers will measure whether IXIUM TWIN causes less damage to the eye's inner lining (endothelial cells) after surgery.

Who can take part? Adults aged 18 and older who have cataracts and are scheduled for surgery may qualify. Only one eye per participant will be included. Patients must be able to attend follow-up visits and provide informed consent.

What does participation involve? Before surgery, participants will have eye exams to check vision, cell health, corneal thickness, and eye pressure. During surgery, they will randomly receive either IXIUM TWIN or HEALON (neither the patient nor the surgeon will choose). After surgery, follow-up visits at 1 day, 7 days, 30 days, and 90 days will monitor healing, vision improvement, and any side effects.

Potential risks and benefits As with any cataract surgery, there are minor risks, such as temporary increased eye pressure, inflammation, or swelling, but these are rare and usually resolve quickly. The benefits include improved vision after cataract removal. If successful, IXIUM TWIN could offer surgeons another high-quality option for protecting the eye during surgery.

Study timeline Patient enrollment begins in January 2025 and ends in June 2025, with follow-ups completing by September 2025. The full study is expected to conclude in early 2026.

This study is sponsored by LCA Pharmaceutical and will take place at four hospitals in France. Participation is voluntary, and patients can withdraw at any time.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) with cataract (described and coded per WHO classification²⁷)
* One eye per patient enrolled in the clinical investigation (IC)
* Intraocular pressure (IOP) controlled or uncontrolled with treatment
* Cataract extraction via phacoemulsification with implantation of a posterior chamber injectable intraocular lens (IOL) through a small incision
* Signed informed consent from both patient and physician
* Patient capable of understanding the IC procedures and geographically stable
* Patient covered by or eligible for a social security/health insurance system

Exclusion Criteria:

* Patient unable to participate in a clinical investigation (IC)
* Pregnant women or those at risk of pregnancy during the study
* Patient under legal guardianship (tutelle), conservatorship (curatelle), or judicial protection (sauvegarde de justice)
* Patient currently enrolled in another clinical investigation at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of Endothelial Cell Loss between pre- and post-operative periods | 90 days
  The primary outcome measure is the percentage of endothelial cell loss observed between the pre-operative and post-operative periods during cataract surgery using viscoelastic devices (OVDs).
  The study assumes that the percentage of endothelial cell loss after using IXIUM TWIN is not clinically worse than that seen with the comparator HEALON, with a non-inferiority margin set at -15%.

SECONDARY OUTCOMES:
Proportion of patients with intraocular pressure (IOP) ≥30 mmHg | 90 days
  Proportion of patients with intraocular pressure (IOP) ≥30 mmHg at each visit.
Slit-lamp biomicroscopy | 90 days
  Slit-lamp biomicroscopy at each visit:
  Multicriteria evaluation graded (1+ to 4+) per the Standardization of Uveitis Nomenclature (SUN) Working Group classification:
  * Corneal edema: Mild (grade 1+), moderate (grade 2+), severe (grade 3+)
  * Corneal opacity (% surface area): ≤25% (grade 1+), 26-50% (grade 2+), ≥51% (grade 3+)
  * Iritis syndrome: Iris involvement only (grade 1+), iridocyclitis (grade 2+), diffuse anterior chamber (AC) involvement (grade 3+)
  * Inflammatory cells in 1×1 mm field: 6-15 (grade 1+), 16-25 (grade 2+), 26-50 (grade 3+), >50 (grade 4+)
  * Anterior chamber flare: Mild (grade 1+), clear details (grade 2+), hazy details (grade 3+), intense with fibrin (grade 4+)
Pachymetry | 90 days
  Measurement of corneal thickness
Best-corrected visual acuity (BCVA) for distance and near vision | 90 days
  Best-corrected visual acuity (BCVA) for distance and near vision at Day 7, 30, and 90 (uncorrected at Day 1).
Assessment of the viscoelastic device (DM) behavior | Post-op
  Assessment of the viscoelastic device (DM) behavior at each surgical step, distinguishing between the two phases: dispersive and cohesive (Likert scale).
Patient satisfaction assessment regarding the procedure (Likert scale) | 90 days
  Patient satisfaction assessment regarding the procedure (Likert scale). Very satisfying - Satisfying - Acceptable - Insufficient
Assessment of adverse events | 90 days
  Assessment of adverse events at all visits

IPD SHARING:
Plan to Share IPD: No